CLINICAL TRIAL: NCT04040816
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SAP-001 in Gout Patients With Hyperuricemia
Brief Title: Placebo Controlled, Multiple Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SAP-001 in Gout Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanton Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Shanton Pharma Pte. Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SAP001-1-002
Record Dates: First submitted 2019-07-17; First posted 2019-08-01 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose A (Experimental): Dose A SAP-001 versus placebo
  Interventions: Drug: SAP-001
- Dose B (Experimental): Dose B SAP-001 versus placebo
  Interventions: Drug: SAP-001
- Dose C (Experimental): Dose C SAP-001 versus placebo
  Interventions: Drug: SAP-001
- Dose D (allopurinol patients) (Experimental): Dose D SAP-001 versus placebo in gout patients who remain on allopurinol
  Interventions: Drug: SAP-001

INTERVENTIONS:
Drug: SAP-001 — SAP-001 or placebo treatment in a 4:1 randomization ratio

SUMMARY:
This is a Phase II, Multicenter, Randomized, Double-blind, Placebo controlled, Multiple Dose study to evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SAP-001 in Gout Patients with Hyperuricemia.

DETAILED DESCRIPTION:
This multiple dose study will include up to 4 cohorts. Each cohort will be comprised of 15 patients who will be dosed with SAP-001 or placebo once daily (QD) for 28 days. Dose escalation from Cohort 1 to Cohort 2 will occur after preliminary data are partially unblinded and safety data along with PK and PD parameters are analyzed and reviewed. Enrollment in Cohort 3 will begin after the last subject is randomized into Cohort 2.

Prior to starting enrollment into Cohort 4, a complete safety assessment of Cohorts 1, 2 and 3 will be performed to select the dose to be used in Cohort 4.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 and ≤ 75 years of age.
2. Body mass index (BMI) ≥ 19 and ≤ 42 kg/m2 at screening.
3. sUA levels ≥ 7.5 mg/dL during screening and at check-in (Day -1).
4. Patients must meet the American College of Rheumatology scoring criteria for the classification of primary gout (Neogi et al 2015).
5. Patients must be able to take gout flare prophylaxis with colchicine 0.6 mg QD throughout the study as the primary method to prevent disease flare. If colchicine is not tolerated or contraindicated, naproxen 250 mg BID with or without H2 antagonists will be employed as a second line gout flare prophylactic agent. Gout flare prophylaxis will be initiated at the Day -1 visit in patients who are sUA-lowering agent naïve. For patients that discontinue an sUA-lowering agent(s) (ie, washout from current therapy) during the screening period, gout flare prophylaxis should be initiated at the time of discontinuation of the sUA-lowering agent(s).
6. Is a nonsmoker or light smoker (smokes fewer than 10 cigarettes per day).
7. Female patients either will be postmenopausal (female patients who state they are postmenopausal should have had cessation of menses for > 1 year and have serum follicle-stimulating hormone [FSH] levels > 40 mIU/mL and serum estradiol < 20 pg/mL); or surgically sterile (including bilateral tubal ligation, salpingectomy [with or without oophorectomy], surgical hysterectomy, or bilateral oophorectomy [with or without hysterectomy]) for at least 3 months prior to screening; or will agree to use, from the time of check-in (Day -1) until 90 days following the last dose of study drug, the following forms of contraception: double-barrier method, hormonal contraceptives, barrier with spermicide, diaphragm or cervical cap with spermicide, intrauterine device, oral, implantable, or injectable contraceptives, or a sterile sexual partner. All female patients, except those with documented surgical hysterectomy in medical history, will have a negative urine pregnancy test result prior to enrollment in the study.
8. Male patients either will be surgically sterile or agree to use, from the time of check-in (Day -1) until 90 days following the last dose of study drug, the following forms of contraception: male condom with spermicide and a female partner who is sterile or agrees to use hormonal contraceptives, female condom with spermicide, diaphragm or cervical cap with spermicide, intrauterine device, oral, implantable, or injectable contraceptives. Male patients will refrain from sperm donation from the time of check-in (Day -1) until 90 days following the last dose of study drug.
9. Is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements.

   Cohorts 1 through 3:
10. Patients who are not taking any UA-lowering medications within 2 weeks prior to the dose of study drug. Patients may discontinue sUA-lowering agents (ie, washout from current therapy) during the screening period. In the cases of a patient who must discontinue sUA-lowering agents or a patient not previously taking sUA-lowering agents during the screening period, gout flare prophylaxis should be initiated with colchicine 0.6 mg QD as the primary method to prevent disease flare and be continued during the study period. If colchicine is not tolerated or contraindicated, naproxen 250 mg BID with or without H2 antagonists will be employed as a second line gout flare prophylactic agent.

    Cohort 4:
11. Patient has been on a stable dose of allopurinol as existing urate-lowering therapy for at least 3 months prior to Day 1.

Exclusion Criteria:

1. Female patient is pregnant, planning to get pregnant, or lactating/breastfeeding.
2. Has a history or presence of CS cardiovascular, renal, pulmonary, hepatic, gallbladder or biliary tract, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, which in the investigator's opinion would not be suitable for the study.
3. Serum creatinine level > 1.5 mg/dL and/or estimated glomerular filtration rate (eGFR) ≤ 60 mL/min/1.73 m2 calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (Levey et al 2009; National Institute of Diabetes and Digestive and Kidney Diseases, Estimating Glomerular Filtration Rate) at screening.
4. History of stomach or intestinal surgery (except cholecystectomy, appendectomy, and/or hernia repair will be allowed).
5. History of prescription drug abuse, illicit drug use, or alcohol abuse according to medical history within 6 months prior to the screening visit or any alcohol use for at least 48 hours prior to dosing on Day 1.
6. Positive test for human immunodeficiency virus (HIV).
7. Positive test for hepatitis B virus or hepatitis C virus (HCV) consistent with current infection. Confirmatory tests will be allowed at the discretion of the investigator to rule out false positives.
8. Clinically significant abnormal liver function test at screening or check-in (Day -1), defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 × upper limit of normal (ULN) or total bilirubin > ULN; or a history of CS acute or chronic hepatitis (including infectious, metabolic, autoimmune, genetic, ischemic, or other forms), hepatocirrhosis, or hepatic tumors.
9. Positive screen for alcohol or drugs of abuse (except for patients with a positive drug screen if it is a result of a prescribed medication from their physician) at screening or check-in (Day -1).
10. History of a gout flare that is resolved within 14 days prior to the first dose of study drug on Day 1 (exclusive of chronic synovitis/arthritis). If a gout flare occurs during screening, patients may be rescreened after a period of at least 14 days has passed following the flare.
11. Has a known hypersensitivity to URAT1 inhibitors, XOIs, or related compounds.
12. Receipt of any other investigational product within 30 days prior to the first dose of study drug on Day 1 or planning to take an investigational agent during the study.
13. Use of drugs or nutrients known to significantly modulate cytochrome P450 (CYP)3A activity starting from 14 days prior to the first dose of study drug on Day 1 until EOS (any strong or moderate inhibitors or inducers of CYP3A4, including but not limited to the following: inhibitors such as ketoconazole, miconazole, itraconazole, fluconazole, atazanavir, erythromycin, clarithromycin, ranitidine, cimetidine, verapamil, and diltiazem; and inducers such as rifampicin, rifabutin, glucocorticoids, carbamazepine, phenytoin, phenobarbital, and St. John's wort).
14. Participated in strenuous exercise from 48 hours prior to check-in (Day -1) or during the study through EOS.
15. Has donated or lost a significant volume (> 500 mL) of blood or plasma within 30 days prior to check-in (Day -1).
16. Malignancy within 5 years prior to the screening visit (excluding basal cell carcinoma).
17. Has problems understanding the protocol requirements, instructions, study-related restrictions, and/or problems understanding the nature, scope, and potential consequences of participating in this clinical study.
18. Is unlikely to comply with the protocol requirements, instructions, and/or study-related restrictions (eg, uncooperative attitude, unavailable for follow up, and/or improbability of completing the clinical study).

    Cohorts 1 through 3:
19. Concomitant use of or treatment with any prescription drugs, herbal products, vitamins, minerals, and over-the-counter (OTC) medications that are known to lower sUA levels (eg, allopurinol, febuxistat, probenecid, lesinurad, and peglodicase) within 14 days prior to check-in (Day -1). Exceptions may be made on a case-by-case basis (such as chronic use of low dose aspirin) following discussion and agreement between the investigator and sponsor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days
  Assess the safety and tolerability of multiple ascending doses of oral SAP-001 over 28 days compared to placebo
Cmax | 28 days
  Maximum observed plasma concentration
tmax | 28 days
  Time to maximum observed plasma concentration
AUC0-t | 28 days
  Area under the plasma concentration-time curve from time 0 to time t
AUC0-24h | 28 days
  Area under the plasma concentration-time curve from time 0 until 24 hours postdose
AUC0-∞ | 28 days
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity
λz | 28 days
  Apparent terminal elimination rate constant
t½ | 28 days
  Terminal elimination phase half-life
CL/F | 28 days
  Total body clearance
Vz/F | 28 days
  Volume of distribution
sUA | 28 days
  Serum urate concentration, change from baseline, and percent change from baseline
Creatinine | 28 days
  Creatinine levels, change from baseline, and percent change from baseline

SECONDARY OUTCOMES:
Urate Lowering Effect | 28 days
  Assess the urate lowering effects of serum urate levels at various time points for multiple ascending doses of SAP-001 over 28 days compared to placebo
Inflammation markers including cytokines IL-1β, IL-6, IL-8, and TNFα | 28 days
  Assess the effects of multiple ascending doses of SAP-001 on selected inflammation markers over 28 days compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Celina Cabale-Scholl, DPT, RN, Study Chair — Shanton Pharma
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Anaheim Clinical Trials (ACT), Anaheim, California
  - Miami Research Associates, South Miami, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Vince & Associates Clinical Research, Inc., Overland Park, Kansas
  - M3 Wake Research, Inc, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided